CLINICAL TRIAL: NCT06104020
Title: Randomized Controlled Trial of Lung Ultrasound-Guided Intraoperative Fluid Management Strategies: Assessing Their Impact on Post-operative Pulmonary Complications and Hemodynamics in Shoulder Arthroscopic Surgerys
Brief Title: Lung Ultrasound-Guided Intraoperative Fluid Management Strategies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aia Abdelhameed mohamed mohamed, Resident physician, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: assiut_ICU2012
Record Dates: First submitted 2023-10-08; First posted 2023-10-27 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Shoulder Arthropathy Associated With Other Conditions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Restrictive fluid group (RG) (Active Comparator): The restrictive fluid group (RG) aims to achieve a net zero fluid balance and involves a 2 mL/kg bolus at anesthesia induction, followed by an intraoperative crystalloid infusion at a rate of 4 mL/kg/hr.
  Interventions: Other: Intraoperative fluid management stratigies.
- liberal group (LG) (Active Comparator): The liberal group (LG) will receive a 10 mL/kg bolus at anesthesia induction, followed by an intraoperative crystalloid infusion at a rate of 8 mL/kg/hr [12, 13].
  Interventions: Other: Intraoperative fluid management stratigies.

INTERVENTIONS:
Other: Intraoperative fluid management stratigies. — Regimens of different intraoperative fluid management The restrictive fluid group (RG) aims to achieve a net zero fluid balance and involves a 2 mL/kg bolus at anesthesia induction, followed by an intraoperative crystalloid infusion at a rate of 4 mL/kg/hr.
  The other group of patients, the liberal group (LG), will receive a 10 ml/kg bolus at anesthesia induction,followed by an intraoperative crystalloid infusion at a rate of 8 ml/kg/hr.

SUMMARY:
The primary aim of our study is to leverage lung ultrasound to assess and identify postoperative pulmonary complications following shoulder arthroscopic surgery and the implications of the used irrigation fluid.the investigators will further investigate the impact of intraoperative fluid management strategies on these Postoperative pulmonary complications and their effects on hemodynamics. By harnessing the potential of lung ultrasound in this context, we aspire to enhance both the diagnostic capabilities and overall safety of shoulder arthroscopic surgery, ultimately improving patient outcomes.

DETAILED DESCRIPTION:
Shoulder arthroscopy, a minimally invasive surgical technique, has become a preferred method for addressing conditions like rotator cuff tears and recurrent joint instability due to its advantages, such as reduced post-operative pain and quicker rehabilitation. However, recent attention has shifted to potential complications, including issues related to irrigation fluid, patient positioning in the beach-chair posture, and anesthesia protocols. One key concern is the use of pressurized irrigation fluid, which, while essential for visualization, carries the risk of complications, including subcutaneous emphysema, pneumomediastinum, tension pneumothorax, air embolism, pulmonary edema, and atelectasis. These complications can have systemic effects, emphasizing the need for precise intraoperative fluid management.

Intraoperative fluid management strategies are a subject of continuous debate in the field of surgery, giving rise to three main strategies: 'liberal,' 'restricted,' and 'goal-directed' fluid therapy. These strategies vary in terms of the type of fluid used, timing of administration, and volume administered. While administering large volumes of fluids may improve organ perfusion, it may also increase the incidence of perioperative cardiopulmonary complications. Conversely, fluid restriction may reduce the length of hospital stay but increase the risk of postoperative acute kidney injury. Goal-directed therapy, which tailors fluid administration based on reproducible endpoints, has been associated with improved perioperative outcomes. The Bezold-Jarisch reflex is a cardiovascular reflex that can result in severe bradycardia and vasodilation when activated, especially in fasting patients with beach-chair position and other positions that lead to pooling of the blood in the lower limb and, in turn, lead to a decrease in venous return.

Understanding the intricate relationship between this reflex and intraoperative fluid management is paramount for improving patient safety and surgical outcomes. This reflex can be triggered by various factors, including rapid fluid administration and alterations in venous return, particularly in patients positioned in the beach chair posture.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective shoulder arthroscopic surgery.
* Adults aged 18 years and above.
* Capable of providing informed consent voluntarily.
* No known allergies or sensitivities to substances commonly used in the surgical procedure or study.
* Stable baseline hemodynamics during preoperative evaluation

Exclusion Criteria:

* Patients scheduled for open shoulder surgery.
* Medical Comorbidities:

  * Pulmonary diseases, including chronic pulmonary diseases or pulmonary edema.
  * Previous cardiac diseases such as heart failure, myocardial infarction (MI), hypertension, and known types of arrhythmia.
* Severe Organ Disease: Severe liver or kidney disease.
* Body mass index (BMI) ≥ 35 kg/m².
* Abnormal coagulation function.
* Pregnancy
* Refusal to Participate or Patients who cannot provide informed consent due to cognitive impairment or other reasons.
* Previous shoulder arthroscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
lung ultrasound score (LUS) | 1-One hour before the start of Surgery. 2-Two hours after the End of surgery.
  we will Identify postoperative pulmonary complications using the lung ultrasound score (LUS) following shoulder arthroscopic surgery to assess the implications of the used irrigation fluid and The intraoperative Fluid infusion
  * 0 = normal lung aeration,
  * 1 = moderate loss of aeration
  * 2 = severe loss of aeration
  * 3 = complete loss of lung aeration

SECONDARY OUTCOMES:
Blood Pressure | Continuous recording every 15 minutes from the start of the operation until its end, assessed up to the completion of the surgical procedure.
  Measured in millimeters of Mercury (mm Hg).
Heart Rate | Continuous recording every 15 minutes from the start of the operation until its end, assessed up to the completion of the surgical procedure.
  Measured in Beats per Minute (bpm).
Oxygen Saturation | Continuous recording every 15 minutes from the start of the operation until its end, assessed up to the completion of the surgical procedure.
  Measured in Percentage (%).
Vasopressor Used and Dose | Continuous recording every 15 minutes from the start of the operation until its end, assessed up to the completion of the surgical procedure.
  Measured in milligrams (mg).
Interval for Repeated Dose of the Vasopressor. | Continuous recording every 15 minutes from the start of the operation until its end, assessed up to the completion of the surgical procedure.
  Measured in minutes.
Duration of Action of used Vasopressor | Continuous recording every 15 minutes from the start of the operation until its end, assessed up to the completion of the surgical procedure.
  Measured in Minutes.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Myles PS, Bellomo R, Corcoran T, Forbes A, Peyton P, Story D, Christophi C, Leslie K, McGuinness S, Parke R, Serpell J, Chan MTV, Painter T, McCluskey S, Minto G, Wallace S; Australian and New Zealand College of Anaesthetists Clinical Trials Network and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Restrictive versus Liberal Fluid Therapy for Major Abdominal Surgery. N Engl J Med. 2018 Jun 14;378(24):2263-2274. doi: 10.1056/NEJMoa1801601. Epub 2018 May 9. PMID 29742967
- [Background] Bhaskar SB, Manjuladevi M. Shoulder arthroscopy and complications: Can we afford to relax? Indian J Anaesth. 2015 Jun;59(6):335-7. doi: 10.4103/0019-5049.158729. No abstract available. PMID 26195827
- [Background] Bouhemad B, Mongodi S, Via G, Rouquette I. Ultrasound for "lung monitoring" of ventilated patients. Anesthesiology. 2015 Feb;122(2):437-47. doi: 10.1097/ALN.0000000000000558. No abstract available. PMID 25501898
- [Background] Orebaugh SL. Life-threatening airway edema resulting from prolonged shoulder arthroscopy. Anesthesiology. 2003 Dec;99(6):1456-8. doi: 10.1097/00000542-200312000-00034. No abstract available. PMID 14639165
- [Background] Rains DD, Rooke GA, Wahl CJ. Pathomechanisms and complications related to patient positioning and anesthesia during shoulder arthroscopy. Arthroscopy. 2011 Apr;27(4):532-41. doi: 10.1016/j.arthro.2010.09.008. Epub 2010 Dec 24. PMID 21186092
- [Background] Saeki N, Kawamoto M. Tracheal obstruction caused by fluid extravasation during shoulder arthroscopy. Anaesth Intensive Care. 2011 Mar;39(2):317-8. No abstract available. PMID 21485693
- [Background] Manjuladevi M, Gupta S, Upadhyaya KV, Kutappa AM. Postoperative airway compromise in shoulder arthroscopy: A case series. Indian J Anaesth. 2013 Jan;57(1):52-5. doi: 10.4103/0019-5049.108563. PMID 23716767
- [Background] Jirativanont T, Tritrakarn TD. Upper airway obstruction following arthroscopic rotator cuff repair due to excess irrigation fluid. Anaesth Intensive Care. 2010 Sep;38(5):957-8. No abstract available. PMID 20872997
- [Background] Lee HC, Dewan N, Crosby L. Subcutaneous emphysema, pneumomediastinum, and potentially life-threatening tension pneumothorax. Pulmonary complications from arthroscopic shoulder decompression. Chest. 1992 May;101(5):1265-7. doi: 10.1378/chest.101.5.1265. PMID 1582282
- [Background] Ichai C, Ciais JF, Roussel LJ, Levraut J, Candito M, Boileau P, Grimaud D. Intravascular absorption of glycine irrigating solution during shoulder arthroscopy: a case report and follow-up study. Anesthesiology. 1996 Dec;85(6):1481-5. doi: 10.1097/00000542-199612000-00031. No abstract available. PMID 8968197
- [Background] Bundgaard-Nielsen M, Secher NH, Kehlet H. 'Liberal' vs. 'restrictive' perioperative fluid therapy--a critical assessment of the evidence. Acta Anaesthesiol Scand. 2009 Aug;53(7):843-51. doi: 10.1111/j.1399-6576.2009.02029.x. Epub 2009 Jun 10. PMID 19519723
- [Background] Prowle JR, Chua HR, Bagshaw SM, Bellomo R. Clinical review: Volume of fluid resuscitation and the incidence of acute kidney injury - a systematic review. Crit Care. 2012 Aug 7;16(4):230. doi: 10.1186/cc11345. PMID 22866958
- [Background] Brandstrup B, Tonnesen H, Beier-Holgersen R, Hjortso E, Ording H, Lindorff-Larsen K, Rasmussen MS, Lanng C, Wallin L, Iversen LH, Gramkow CS, Okholm M, Blemmer T, Svendsen PE, Rottensten HH, Thage B, Riis J, Jeppesen IS, Teilum D, Christensen AM, Graungaard B, Pott F; Danish Study Group on Perioperative Fluid Therapy. Effects of intravenous fluid restriction on postoperative complications: comparison of two perioperative fluid regimens: a randomized assessor-blinded multicenter trial. Ann Surg. 2003 Nov;238(5):641-8. doi: 10.1097/01.sla.0000094387.50865.23. PMID 14578723
- [Background] Kinsella SM, Tuckey JP. Perioperative bradycardia and asystole: relationship to vasovagal syncope and the Bezold-Jarisch reflex. Br J Anaesth. 2001 Jun;86(6):859-68. doi: 10.1093/bja/86.6.859. PMID 11573596
- [Background] D'Alessio JG, Weller RS, Rosenblum M. Activation of the Bezold-Jarisch reflex in the sitting position for shoulder arthroscopy using interscalene block. Anesth Analg. 1995 Jun;80(6):1158-62. doi: 10.1097/00000539-199506000-00016. PMID 7762845
- [Background] Myles P, Bellomo R, Corcoran T, Forbes A, Wallace S, Peyton P, Christophi C, Story D, Leslie K, Serpell J, McGuinness S, Parke R; Australian and New Zealand College of Anaesthetists Clinical Trials Network, and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Restrictive versus liberal fluid therapy in major abdominal surgery (RELIEF): rationale and design for a multicentre randomised trial. BMJ Open. 2017 Mar 3;7(3):e015358. doi: 10.1136/bmjopen-2016-015358. PMID 28259855
- [Background] Mongodi S, Bouhemad B, Orlando A, Stella A, Tavazzi G, Via G, Iotti GA, Braschi A, Mojoli F. Modified Lung Ultrasound Score for Assessing and Monitoring Pulmonary Aeration. Ultraschall Med. 2017 Oct;38(5):530-537. doi: 10.1055/s-0042-120260. Epub 2017 Mar 14. PMID 28291991